CLINICAL TRIAL: NCT05782322
Title: Effects and Neural Mechanisms of Training Involving Rhythmic Auditory Stimulation on Upper-limb Movements in Patients With Parkinson's Disease
Brief Title: Effects and Mechanisms of RAS Training on Upper-limb Movements in PD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, FAN Wei, PhD Student, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HongKongPU21037721r_20230221
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Acoustic Stimulation; Parkinson Disease; Electroencephalography
Keywords: Acoustic Stimulation; Parkinson Disease; Movement; Electroencephalography
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PD-RAS (Experimental): training involving RAS
  Interventions: Behavioral: Upper-limb training involving RAS
- PD-noRAS (Active Comparator): training without the aid of RAS
  Interventions: Behavioral: Upper-limb training without the aid of RAS
- HC-RAS (Experimental): training involving RAS
  Interventions: Behavioral: Upper-limb training involving RAS
- HC-noRAS (Active Comparator): training without the aid of RAS
  Interventions: Behavioral: Upper-limb training without the aid of RAS

INTERVENTIONS:
Behavioral: Upper-limb training involving RAS — Three target bowls, labeled as the left, middle, and right target bowl, will be placed on the table at an equal distance from the main bowl. The distance between a target bowl and the main bowl is set at 30 cm. Wooden beads with a diameter of 2 cm will be put in target bowls. The main bowl will be placed in front of the patient.
  Patients will be asked to listen to the RAS sound, use the right hand to take one bead at a time from the left target bowl to the main bowl, repeat this movement for the middle and right target bowls, and keep repeating this order. They should keep their movements consistent with the sound of the RAS, with one RAS sound corresponding to one pick-up movement.
  Each daily training will consist of three rounds separated by two 5-minute breaks. Each round will consist of four consecutive sessions (for each session: 2-minute training followed by a 30-second break). The training will last for a total of 7 days.
  Arms: HC-RAS; PD-RAS
Behavioral: Upper-limb training without the aid of RAS — Three target bowls, labeled as the left, middle, and right target bowl, will be placed on the table at an equal distance from the main bowl. The distance between a target bowl and the main bowl is set at 30 cm. Wooden beads with a diameter of 2 cm will be put in target bowls. The main bowl will be placed in front of the patient.
  Patients will be asked to use the right hand to take one bead at a time from the left target bowl to the main bowl, repeat this movement for the middle and right target bowls, and keep repeating this order. They are asked to execute the task as fast as possible.
  Each daily training will consist of three rounds separated by two 5-minute breaks. Each round will consist of four consecutive sessions (for each session: 2-minute training followed by a 30-second break). The training will last for a total of 7 days.
  Arms: HC-noRAS; PD-noRAS

SUMMARY:
Introduction Bradykinesia (i.e., slow movements) is one of the most prominent symptoms of Parkinson's disease (PD) and has a negative impact on quality of life. Rhythmic auditory stimulation (RAS), a widely used and promising treatment technique, has been shown to effectively improve gait speed in PD patients. However, only few studies have explored effects and neural mechanisms of RAS on upper-limb movements. We will conduct two studies to investigate effects and mechanisms of RAS on upper-limb movements in PD patients. The purpose of this study is to examine effects and neural mechanisms of upper-limb movement training involving RAS in PD patients.

Methods This study will recruit patients with PD and healthy controls. This study will randomly assign PD patients into two groups: the PD-RAS group and the PD-noRAS group, and healthy controls into the HC-RAS group and the HC-noRAS group. A 7-day upper-limb training involving RAS (for the PD-RAS group and the HC-RAS group) or without RAS (for the PD-noRAS group and the HC-noRAS group) will be provided. EEG and behavioral assessments will be conducted before and after the first day of training, and after the seven-day training program. Two-way repeated measures analysis of variance will be performed to investigate the group and time effects on upper-limb function and neural activity.

Study significance The training program will serve as a reference for clinical practitioners who are interested in using RAS in clinical training for PD patients.

ELIGIBILITY:
Inclusion Criteria:

* (a) idiopathic PD diagnosed by a neurologist based on the Movement Disorders Society clinical diagnostic criteria;
* (b) the Hoehn and Yahr stage is 2 or 3, meaning that bilateral movement problems or combination with mild postural instability;
* (c) a score of Montreal Cognitive Assessment (MoCA) is equal to or higher than 21 to ensure that they understand experimental instructions;
* (d) a score of Edinburgh Handedness Inventory is above 60 to ensure that they are right-handed;
* (e) types and doses of medications remain unchanged in the past month right before participation.
* Age- and sex-matched healthy controls who filled the criteria (c) and (d) will be recruited from communities.

Exclusion Criteria:

* the presence of medical conditions or diseases that may affect hand movements, vision, or hearing based on self-report.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | Assessments will be performed before the first day of training.
  The power (unit:Watt) of EEG will be calculated.
Electroencephalography (EEG) | Assessments will be performed after the seven-day training program.
  The power (unit:Watt) of EEG will be calculated.
Electroencephalography (EEG) | Assessments will be performed before the first day of training.
  The functional connectivity (unit:coherence) of EEG will be calculated.
Electroencephalography (EEG) | Assessments will be performed after the seven-day training program.
  The functional connectivity (unit:coherence) of EEG will be calculated.
The box and block test (BBT) | Assessments will be performed before the first day of training.
  The BBT is used to measure gross manual dexterity as well as upper-limb movement speed.
The box and block test (BBT) | Assessments will be performed after the seven-day training program.
  The BBT is used to measure gross manual dexterity as well as upper-limb movement speed.
The nine hole peg test (NHPT) | Assessments will be performed before the first day of training.
  The NHPT is a widely used measure of hand dexterity in a broad range of ages and populations.
The nine hole peg test (NHPT) | Assessments will be performed after the seven-day training program.
  The NHPT is a widely used measure of hand dexterity in a broad range of ages and populations.

SECONDARY OUTCOMES:
The Jebsen Hand Function Test (JHFT) | Assessments will be performed before the first day of training.
  The Jebsen Hand Function Test (JHFT) evaluated unimanual performance in activities of daily living through six standardized tasks: card turning, small object manipulation, simulated feeding, checker stacking, and moving both light and heavy objects. We modified the original seven-item test by excluding the writing task to accommodate Chinese-speaking participants, following established protocols for cross-cultural adaptation. Performance was measured by completion time for each task, with shorter times indicating better hand function. The JHFT demonstrates excellent test-retest reliability in PD patients (intraclass correlation coefficients: 0.89-0.97).
The Jebsen Hand Function Test (JHFT) | Assessments will be performed after the 7-day training.
  The Jebsen Hand Function Test (JHFT) evaluated unimanual performance in activities of daily living through six standardized tasks: card turning, small object manipulation, simulated feeding, checker stacking, and moving both light and heavy objects. We modified the original seven-item test by excluding the writing task to accommodate Chinese-speaking participants, following established protocols for cross-cultural adaptation. Performance was measured by completion time for each task, with shorter times indicating better hand function. The JHFT demonstrates excellent test-retest reliability in PD patients (intraclass correlation coefficients: 0.89-0.97).
Ruler Drop Test (RDT) | Assessments will be performed before the first day of training.
  We assessed reaction time using the Ruler Drop Test (RDT). During this test, a ruler was positioned vertically between the participant's thumb and index finger, with its zero mark aligned at the fingertips. Following a ready signal from the participant, the examiner released the ruler without warning, requiring the participant to catch it as quickly as possible upon visual detection of movement. The falling distance was recorded, with greater distances indicating longer reaction times. The test was repeated three times, and the average distance was calculated. This measure reflects neuromotor processing speed, encompassing both visual information processing and movement initiation time.
Ruler Drop Test (RDT) | Assessments will be performed after the 7-day training.
  We assessed reaction time using the Ruler Drop Test (RDT). During this test, a ruler was positioned vertically between the participant's thumb and index finger, with its zero mark aligned at the fingertips. Following a ready signal from the participant, the examiner released the ruler without warning, requiring the participant to catch it as quickly as possible upon visual detection of movement. The falling distance was recorded, with greater distances indicating longer reaction times. The test was repeated three times, and the average distance was calculated. This measure reflects neuromotor processing speed, encompassing both visual information processing and movement initiation time.

CONTACTS AND LOCATIONS:
Overall Officials: Wei FAN (PhD student), MSc, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bengtsson SL, Ullen F, Ehrsson HH, Hashimoto T, Kito T, Naito E, Forssberg H, Sadato N. Listening to rhythms activates motor and premotor cortices. Cortex. 2009 Jan;45(1):62-71. doi: 10.1016/j.cortex.2008.07.002. Epub 2008 Oct 30. PMID 19041965
- [Background] Braunlich K, Seger CA, Jentink KG, Buard I, Kluger BM, Thaut MH. Rhythmic auditory cues shape neural network recruitment in Parkinson's disease during repetitive motor behavior. Eur J Neurosci. 2019 Mar;49(6):849-858. doi: 10.1111/ejn.14227. Epub 2018 Dec 3. PMID 30375083
- [Background] Buard I, Dewispelaere WB, Thaut M, Kluger BM. Preliminary Neurophysiological Evidence of Altered Cortical Activity and Connectivity With Neurologic Music Therapy in Parkinson's Disease. Front Neurosci. 2019 Feb 19;13:105. doi: 10.3389/fnins.2019.00105. eCollection 2019. PMID 30837830
- [Background] Cahn DA, Sullivan EV, Shear PK, Pfefferbaum A, Heit G, Silverberg G. Differential contributions of cognitive and motor component processes to physical and instrumental activities of daily living in Parkinson's disease. Arch Clin Neuropsychol. 1998 Oct;13(7):575-83. PMID 14590618
- [Background] Chen JL, Penhune VB, Zatorre RJ. Listening to musical rhythms recruits motor regions of the brain. Cereb Cortex. 2008 Dec;18(12):2844-54. doi: 10.1093/cercor/bhn042. Epub 2008 Apr 3. PMID 18388350
- [Background] Dalrymple-Alford JC, MacAskill MR, Nakas CT, Livingston L, Graham C, Crucian GP, Melzer TR, Kirwan J, Keenan R, Wells S, Porter RJ, Watts R, Anderson TJ. The MoCA: well-suited screen for cognitive impairment in Parkinson disease. Neurology. 2010 Nov 9;75(19):1717-25. doi: 10.1212/WNL.0b013e3181fc29c9. PMID 21060094
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E, Mercier L. Validation of the Box and Block Test as a measure of dexterity of elderly people: reliability, validity, and norms studies. Arch Phys Med Rehabil. 1994 Jul;75(7):751-5. PMID 8024419
- [Background] Dong VA, Fong KN, Chen YF, Tseng SS, Wong LM. 'Remind-to-move' treatment versus constraint-induced movement therapy for children with hemiplegic cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2017 Feb;59(2):160-167. doi: 10.1111/dmcn.13216. Epub 2016 Aug 9. PMID 27503605
- [Background] Fan W, Li J, Wei W, Xiao SH, Liao ZJ, Wang SM, Fong KNK. Effects of rhythmic auditory stimulation on upper-limb movements in patients with Parkinson's disease. Parkinsonism Relat Disord. 2022 Aug;101:27-30. doi: 10.1016/j.parkreldis.2022.06.020. Epub 2022 Jun 23. PMID 35763906
- [Background] Ghai S, Ghai I, Schmitz G, Effenberg AO. Effect of rhythmic auditory cueing on parkinsonian gait: A systematic review and meta-analysis. Sci Rep. 2018 Jan 11;8(1):506. doi: 10.1038/s41598-017-16232-5. PMID 29323122
- [Background] Koshimori Y, Thaut MH. Future perspectives on neural mechanisms underlying rhythm and music based neurorehabilitation in Parkinson's disease. Ageing Res Rev. 2018 Nov;47:133-139. doi: 10.1016/j.arr.2018.07.001. Epub 2018 Jul 10. PMID 30005957
- [Background] Leuk JSP, Low LLN, Teo WP. An Overview of Acoustic-Based Interventions to Improve Motor Symptoms in Parkinson's Disease. Front Aging Neurosci. 2020 Aug 14;12:243. doi: 10.3389/fnagi.2020.00243. eCollection 2020. PMID 32922283
- [Background] Thaut MH, McIntosh GC, Rice RR, Miller RA, Rathbun J, Brault JM. Rhythmic auditory stimulation in gait training for Parkinson's disease patients. Mov Disord. 1996 Mar;11(2):193-200. doi: 10.1002/mds.870110213. PMID 8684391
- [Background] Wang SM, Chan ST, Wong YL, Hsu HM, Lee CY, Check CY, Leung CK. Rhythmic auditory stimulation incorporated in training improved movements in individuals with psychotic-like experiences. Eur Arch Psychiatry Clin Neurosci. 2023 Jun;273(4):995-1005. doi: 10.1007/s00406-022-01524-3. Epub 2022 Nov 24. PMID 36422679